CLINICAL TRIAL: NCT05520931
Title: Pain-related Long Covid in Covid-19 Survivors
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Brian Duborg Ebbesen, PhD fellow, Aalborg University
Other Study IDs: 2021-056227
Record Dates: First submitted 2022-08-29; First posted 2022-08-30 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; Pain, Chronic
Keywords: Covid-19; Coronavirus; Chronic Pain; Persistant pain; Long Covid; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Chronic Pain; Coronavirus Infections; Post-Acute COVID-19 Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalization group: Previously hospitalized Covid-19 survivors who have been admittet to the hospital with or because of SARS-CoV-2 infection. Time from infection date start is > 6 months. The group is anticipated to encompass 2.182 privously hospitalized adult patients.
  Interventions: Other: Questionnaire and register-based data assessment
- PCR+ group: Non-hospitalized Covid-19 survivors that has previously testet positive in an Polymerase chain reaction test without being admittet to the hospital. Time from infection data start is > 6 months. The group will include almost the total population of adults who have tested positive in a Polymerase Chain Reaction test. Those with secret adresses and those without access to digital mail (information channel of the questionnaire) will be excluded being approcimatelyh 7% of 650.000 possible participants. The group encompasses 593.741 participants.
  Interventions: Other: Questionnaire and register-based data assessment

INTERVENTIONS:
Other: Questionnaire and register-based data assessment — Primary data will be collected via a generic questionnaire from the two groups. Secondary data will consist of register-based socio-economic data and medical charts data collected from the Danish Health Data Authority and Denmark' Statistics.

SUMMARY:
The exploratory project aims to investigate the presence of pain as a long Covid-19 symptom in previously hospitalised patients and in non-hospitalised persons previously tested positive in a PCR test.

DETAILED DESCRIPTION:
The main objectives investigated will be to determine the general prevalence of pain symptoms In Covid-19 survivors, correlating and analysing the role of previously comorbidities in the development of pain symptom in Covid-19 survivors, and to understand the prevalence of pain related long Covid-19 symptoms for future characterisations. Hence, the projects main outcome will be to try to understand why som Covid-19 survivors develop persistant pain and others don't. Furthermore, the project plan to analyse gender and age differences, and data between Covid-19 waves as well as any possible association between pain prevalence and time after positive PCR-test.

ELIGIBILITY:
Inclusion Criteria:

* Previously infected with SARS-CoV-2 virus

Exclusion Criteria:

* Participants under the age of 18
* Hidden/secret address/name
* No access to digital mail (the channel of data collection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital group: All patients aged 18 or above that has been admittet to a hospitals in Denmark between 1st of Mach 2020 and 31st of December 2021.
  PCR+ group: All persons aged 18 or above that between 1st March 2020 and 31st of December 2021 have tested positive in a PCR test without hospital admission.
Sampling Method: Non-Probability Sample
Enrollment: 600000 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Persistent pain in Covid-19 survivors | Above six months after a SARS-CoV-2 infection
  Detection of possible differences in Covid-19 survivors with or without persistent pain after a SARS-CoV-2 infection as collected via questionnaire data

SECONDARY OUTCOMES:
The role of comorbidities in the development of persistent pain in Covid-19 survivors | Above six months after a SARS-CoV-2 infection
  Register-based medical charts from hospitalization correlated with self-reported pain from the questionnaire data
The role of comorbidities in the development of persistent pain in Covid-19 survivors II | Above six months after a SARS-CoV-2 infection
  Register-based data about positive PCR-test correlated with self-reported pain from the questionnaire data
The role of socio-economic impact on the development of persistent pain in Covid-19 survivors | Above six months after a SARS-CoV-2 infection
  Register-based data of socio-economic variables that could influence self-rated perception of pain

CONTACTS AND LOCATIONS:
Overall Officials: Lars Arendt-Nielsen, Dr.med, PhD, Study Director — North Denmark Region; Brian D Ebbesen, PhD student, Principal Investigator — North Denmark Region
Locations (1):
- The North Denmark Region, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided